CLINICAL TRIAL: NCT05966467
Title: A Long-Term, Prospective, Observational, Registry of Patients With Anti-Aquaporin 4 Antibody-Positive (AQP4+) Neuromyelitis Optica Spectrum Disorder (NMOSD) Treated With Alexion Complement Component 5 (C5) Inhibitor Therapies (ALXN-C5IT)
Brief Title: Registry of Patients With AQP4+ NMOSD Treated With Alexion C5 Inhibitor Therapies
Status: Recruiting | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: D9282C00003
Record Dates: First submitted 2023-07-07; First posted 2023-07-28 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Neuromyelitis Optica Spectrum Disorder; NMOSD; AQP4+ NMOSD
Keywords: Neuromyelitis Optica Spectrum Disorder; NMOSD; C5 Inhibitor Therapies; AQP4+ NMOSD; Patient Registry; Alexion C5IT; Soliris
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Long-term, multicenter, multinational, observational, registry of patients with AQP4+ NMOSD that is designed to collect data on clinical outcomes and safety in patients prescribed Alexion C5 inhibitor therapies (C5IT). The registry will also collect data on patient reported outcomes (PROs), quality of life (QoL), and targeted AQP4+ NMOSD therapies used to provide evidence on the real-world impact of ALXN-C5IT on patients with AQP4+ NMOSD.

DETAILED DESCRIPTION:
At the time of enrollment in the Registry, participant records will be queried for retrospective information about the participant's medical history and AQP4+ NMOSD treatment history for the time period beginning 1 year prior to ALXN-C5IT initiation through Registry enrollment. The duration of data collection for the Registry will be approximately 5 years from the day the last participant is enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥ 18 years of age at the time of enrollment in the Registry.
* Participant must have a confirmed diagnosis of AQP4+ NMOSD.
* At the time of enrollment in the Registry, participants must be receiving treatment with ALXN-C5IT for the purpose of chronic relapse prevention in a manner consistent with the local label. Specifically, they should have received at least 1 dose of eculizumab within 4 weeks prior to enrollment or at least 1 dose of ravulizumab within 12 weeks prior to enrollment.
* Participants must have both the following historical data available to be enrolled in the Registry: ALXN-C5IT dosing information since initiation and number and types of relapses from 1 year prior to ALXN-C5IT initiation through Registry enrollment.

Exclusion Criteria:

* Participants currently enrolled in an interventional clinical study for the treatment of AQP4+ NMOSD in which the intervention is a drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a diagnosis of AQP4+ NMOSD who are being treated with ALXN-C5IT at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Annualized Relapse Rate (ARR) | Up to approximately 5 years
  The ARR is defined as the total number of relapses divided by the total number of participant-years.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Lopez, Principal Investigator — Hospital Aleman
Locations (25):
- United States (6):
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Research Site, Boston, Massachusetts
  - Clinical Trial Site, Chapel Hill, North Carolina
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Plano, Texas
  - Clinical Trial Site, Milwaukee, Wisconsin
- Clinical Trial Site, Buenos Aires, Argentina
- Clinical Trial Site, Burnaby, British Columbia, Canada
- China (6):
  - Clinical Trial Site, Beijing
  - Clinical Trial Site, Guangzhou
  - Clinical Trial Site, Henan
  - Clinical Trial Site, Shanghai
  - Clinical Trial Site, Sichuan
  - Clinical Trial Site, Wuhan
- Germany (3):
  - Clinical Trial Site, Dresden
  - Clinical Trial Site, Essen
  - Clinical Trial Site, München
- Clinical Trial Site, Naples, Italy
- Japan (4):
  - Clinical Trial Site, Fukuoka
  - Clinical Trial Site, Kawasaki
  - Clinical Trial Site, Miyagi
  - Clinical Trial Site, Tokyo
- South Korea (3):
  - Clinical Trial Site, Daejeon
  - Clinical Trial Site, Gyeonggi-do
  - Clinical Trial Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR